CLINICAL TRIAL: NCT05680701
Title: Understanding and Modulating Cortical Dynamics of Dual-task Standing in Older Adults With Mild Cognitive Impairment
Brief Title: Modulating Cortical Dynamics of Dual-task Standing in MCI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hebrew SeniorLife (Other)
Responsible Party: Principal Investigator, Melike Kahya, Postdoctoral Research Fellow, Hebrew SeniorLife
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: Pro00067596
Record Dates: First submitted 2022-12-19; First posted 2023-01-11 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-01

CONDITIONS: Aging; Mild Cognitive Impairment
Keywords: aging; mild cognitive impairment; non-invasive brain stimulation
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- real tACS (Active Comparator): The investigators will administer the transcranial alternating current stimulation (tACS) intervention at 10 Hz to the participants. This intervention will utilize 6 electrodes; electrode placement and current parameters for each electrode have been optimized using a standard brain to generate an average electric field of 0.25 V/m. To ensure adherence to current safety recommendations for tACS, optimizations will be constrained to a maximum of total injected current 4.0 mA and a max. current per electrode of 2.0 mA. Stimulation will start and end with a 60 s ramp up/down to maximize comfort. This standard approach is both well-tolerated and safe in older adults. In a separate visit, we will use an active sham in which very low-level currents (0.5 mA total) will be transferred between electrodes in close proximity on the scalp throughout the entire 20-minute session.
  Interventions: Other: real tACS
- sham tACS (Sham Comparator): The investigators will administer the sham tACS intervention to the participants. They will use an active sham in which very low-level alternating currents (0.5 mA total) will be transferred between electrodes in close proximity on the scalp throughout the entire 20-minute session.
  Interventions: Other: sham tACS

INTERVENTIONS:
Other: real tACS — The participant will receive one session of 10 Hz tACS for 20-minutes
  Arms: real tACS
Other: sham tACS — The participant will receive one session of active-sham tACS for 20-minutes
  Arms: sham tACS

SUMMARY:
The investigators have designed a brain stimulation study to understand its effect on an individual's standing, walking, and thinking abilities in older adults with and without mild cognitive impairments (MCI). The transcranial alternating current stimulation (tACS) technology has been safely and effectively used in hundreds of individuals. The purpose of this study is to test whether a single session of tACS as compared to sham intervention, improves standing, walking, and thinking in older adults with and without mild cognitive impairments (MCI). Approximately 60 people will take part in this study.

DETAILED DESCRIPTION:
Mild Cognitive Impairment (MCI) represents a common prodromal phase of dementia1. As compared to older adults who are cognitively-intact, those with MCI tend to exhibit poor "dual-task" standing balance performance; that is, the ability to maintain balance when standing and simultaneously performing an unrelated cognitive task. Moreover, those older adults who have worse dual-task standing balance are more likely to suffer falls and develop dementia. As such, strategies designed to understand and enhance the brain functionality involved in dual-task standing balance hold great promise to improve daily life function, and potentially, reduce the risk of dementia in this population.

Surface electroencephalography (EEG) allows non-invasive assessment of brain activity dynamics over short periods of time, even when standing. It has been demonstrated in younger and older adults that dual-task standing is associated with brain activity fluctuations at specific frequencies. A recent study from our laboratory demonstrated that in older adults, 1) performance of a serial subtraction cognitive task when standing reduces fronto-central alpha power (i.e., fluctuations in the 8-13 Hz band), and 2) those with lower fronto-central alpha power when dual tasking exhibit worse dual task standing balance. Intriguingly, numerous studies have separately linked diminished alpha activity with worse performance on executive function and visuomotor tasks, as well as global cognitive decline in older adults. We therefore contend that therapeutic strategies designed to increase alpha activity hold promise to improve dual-task standing performance, and many other cognitive-motor functions in older adults with and without MCI. To date, however, the effects of enhancing fronto-central alpha activity to improve dual-task balance in older adults with and without MCI have not been studied.

Transcranial alternating stimulation (tACS) is a safe, non-invasive brain stimulation technique that utilizes low-amplitude alternating currents to modulate brain activity and entrain specific cortical rhythms depending on the applied stimulation frequency. Targeting alpha band (10 Hz) in the frontal region has been shown to improve cognitive functioning in healthy older adults. However, no studies have investigated the effect of 10 Hz fronto-central stimulation on EEG alpha activity and postural sway outcomes during dual-task standing in older adults with and without MCI. We thus propose to conduct a within-subject cross-over, sham-controlled study in 30 older adults without an overt disease and 30 older adults with MCI. Participants will undergo dual-task standing and cognitive assessments immediately before and after single sessions of 10 Hz tACS (fronto-central alpha stimulation), and active-sham to understand the effect of different stimulation parameters on dual-task standing performance in older adults. We hypothesize that (1) older adults with MCI will demonstrate decreased EEG alpha power during dual-task standing compared to healthy controls, and decreased alpha power will be associated with worse balance outcomes during dual-task standing, and (2) compared to the pre-stimulation condition, participants will exhibit a greater increase in alpha power during the dual-task standing condition following tACS as compared to sham stimulation, and the increase in alpha power from pre-to-post tACS will correlate with a decrease in dual-task postural sway speed from pre-to-post tACS in older adults with and without MCI.

ELIGIBILITY:
Inclusion Criteria:

Healthy older adults:

Our target population will be healthy older men and women who are cognitively intact. We will also ensure that participants are not so impaired that they cannot safely participate nor potentially benefit from the intervention.

* Age 65+ without any cognitive impairment (based in MoCA or TICS)
* Willing and capable to give informed consent for the participation in the study after it has been thoroughly explained able and willing to comply with all study requirements informed consent form was signed
* Ability to stand and walk independently
* Understanding of the informed consent form (ICF) will be assessed by asking the participant to answer the following three questions: 1) What is the purpose of this study? 2) What are the risks of study involvement? 3) If you decide to participate, are you allowed to withdraw from the study at any time? Answers will be recorded by study personnel on the "Assessment of Protocol Understanding" form. Insufficient understanding will be defined by one or more incorrect answers, as determined at the discretion of the investigator.

Older MCI participants:

* Age 65+
* Who have been diagnosed with cognitive impairment (based in MoCA or TICS and Clinical Dementia Rating: CDR 0.5)
* Ability to stand and walk independently
* Willing and capable to give informed consent for the participation in the study after it has been thoroughly explained
* Cut off of MOCA score >18 will be applied
* Able and willing to comply with all study requirements informed consent form was signed
* Understanding of the ICF will be assessed by asking the participant to answer the following three questions: 1) What is the purpose of this study? 2) What are the risks of study involvement? 3) If you decide to participate, are you allowed to withdraw from the study at any time? Answers will be recorded by study personnel on the "Assessment of Protocol Understanding" form (see attached). Insufficient understanding will be defined by one or more incorrect answers, as determined at the discretion of the investigator.

Exclusion Criteria:

Healthy older adults:

Exclusion Criteria have been selected to ensure safety and optimize compliance while minimizing confounds due to overt disease or conditions that may significantly influence study outcomes.

* Potentially eligible individuals will complete the Montreal Cognitive Assessment (MoCA) - score < 26
* Major psychiatric co-morbidity including major depressive disorder, schizophrenia or psychosis
* Self-reported diagnosis of Parkinson's disease, Alzheimer's disease or dementia, multiple sclerosis, history of stroke or other neurodegenerative disorder.
* Self-reported active cancer for which chemo-/radiation therapy is being received.
* Blindness or other disabilities that prevent task performance
* Contraindications to tACS, as recorded on a standardized screening questionnaire, which include a reported seizure within the past two years, use of neuroactive drugs, self-reported presence of specific implanted medical devices (e.g., deep brain stimulator, medication infusion pump, cochlear implant, pacemaker, etc.), or the presence of any active dermatological condition, such as eczema, on the scalp
* Inability to stand or ambulate unassisted for at least 25 feet
* Hospitalization within the past 3 months due to acute illness or as a result of musculoskeletal injury significantly affecting gait and balance

Older MCI participants:

* Cut off of MOCA score <18 will be applied
* Major psychiatric co-morbidity including major depressive disorder, schizophrenia or psychosis
* Blindness or other disabilities that prevent task performance
* Self-reported history of stroke or neurodegenerative disorders other than MCI.
* Self-reported active cancer for which chemo-/radiation therapy is being received.
* Contraindications to tACS, as recorded on a standardized screening questionnaire, which include a reported seizure within the past two years, use of neuro-active drugs, self-reported presence of specific implanted medical devices (e.g., deep brain stimulator, medication infusion pump, cochlear implant, pacemaker, etc.), or the presence of any active dermatological condition, such as eczema, on the scalp.

Ages: 65 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-03-13 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
EEG alpha-band power | Change from immediately before and after each 20-minute session of tACS
  EEG oscillations and frequency coupling at 8-13 Hz
Postural sway speed | Change from immediately before and after each 20-minute session of tACS
  This metric assesses the ability to control standing posture

SECONDARY OUTCOMES:
Timed Up and Go Test (TUG) | This outcome will be assessed immediately before and after each 20-minute session of tACS
  A common field test of mobility
Postural sway area | This outcome will be assessed immediately before and after each 20-minute session of tACS
  This metric assesses the ability to control standing posture
Postural sway path | This outcome will be assessed immediately before and after each 20-minute session of tACS
  This metric assesses the ability to control standing posture
EEG theta-band power | This outcome will be assessed immediately before and after each 20-minute session of tACS
  EEG oscillations and frequency coupling at 4-7 Hz
EEG beta-band power | This outcome will be assessed immediately before and after each 20-minute session of tACS
  EEG oscillations and frequency coupling at 13-30 Hz

CONTACTS AND LOCATIONS:
Overall Officials: Melike Kahya, Principal Investigator — Marcus Institute for Aging Research
Locations (1):
- Marcus Institute for Aging Research, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The HSL Marcus Institute for Aging Research will promote the development of new research and new investigators by making the data available to outside investigators. The database will include demographic, clinical, functional, and neurophysiologic data from all participants.
  All data will be stripped of primary identifiers and entered into a master database. All data collection procedures, variable definitions and codes, field locations, and frequencies will be documented in a separate file.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: The investigators will make the data and associated documentation available once summary data are published or otherwise made available, starting six months after publication.
Access Criteria: The investigators will make the data and associated documentation available to users only under a data-sharing agreement that provides for: 1) a commitment to using data only for research purposes and not to identify any particular participant; 2) a commitment to securing the data using appropriate computer technology; and 3) a commitment to destroying or returning the data after analyses are completed. The availability of data will be advertised over the Internet through websites maintained by Hebrew SeniorLife and Harvard Medical School.
  All investigators wishing to access the data will submit a brief proposal describing their research project, data needs, regulatory approvals, and mechanisms to assure patient confidentiality. Upon affirmative review by the Principal Investigator and co-investigators of this study, a data-sharing agreement will be signed and the requesting investigators will be given a working data file and appropriate documentation.